CLINICAL TRIAL: NCT04997174
Title: Comparison of Postoperative Pain Management in Patients Undergoing Laparoscopic Colorectal Surgery Under Enhanced Recovery After Surgery (ERAS) Program, Laparoscopic Colorectal Surgery Without ERAS and Open Colorectal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Associate Professor, Prince of Songkla University
Other Study IDs: REC.64-290-8-1
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ERAS: Patients undergoing laparoscopic colorectal surgery with ERAS
  Interventions: Drug: Celecoxib
- Non ERAS: Patients undergoing laparoscopic colorectal surgery without ERAS
- Open: Patients undergoing open colorectal surgery

INTERVENTIONS:
Drug: Celecoxib — Patients in ERAS group received celecoxib
  Groups: ERAS

SUMMARY:
This is a retrospective study to compare postoperative pain intensity in patients going laparoscopic colorectal surgery with Enhanced Recovery after Surgery (ERAS), without ERAS and open colorectal surgery.

DETAILED DESCRIPTION:
This study is a matched case-control study. Control patients will be matched to ERAS cases in a 1:1:1 ratio (laparoscopic surgery with ERAS protocol : laparoscopic surgery without ERAS protocol : open surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colorectal surgery under ERAS program and those with the same sort of laparoscopic surgery without ERAS program as well as those with open colorectal surgery with complete required recorded data.

Exclusion Criteria:

* 1. Patients with incomplete required data on record.
* 2. Those with any major intraoperative or postoperative complications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group of interest: Laparoscopic colorectal surgery with Enhanced Recovery after Surgery (ERAS) program defined as patients undergoing laparoscopic colorectal surgery [laparoscopic right / left hemicolectomy, laparoscopic low anterior resection, laparoscopic abdominoperineal resection (APR) and others] under ERAS protocol.
  Control 1: Laparoscopic colorectal surgery without Enhanced Recovery after Surgery (ERAS) program defined as patients undergoing laparoscopic colorectal surgery [laparoscopic right / left hemicolectomy, laparoscopic low anterior resection, laparoscopic abdominoperineal resection (APR) and others] under conventional protocol.
  Control 2: Open colorectal surgery defined as patients undergoing open laparotomy for colorectal surgery [open right / left hemicolectomy, open low anterior resection, open abdominoperineal resection (APR) and others].
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Until discharge (5-7 days)
  Pain score (Verbal Numerical Rating Scale: VNRS) after surgery, VNRS consists of 0-10, where 0 means no pain and 10 means worst pain imaginable

SECONDARY OUTCOMES:
Opioid | Until discharge (5-7 days)
  Amount of postoperative opioid consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Sasikaan Nimmaanrat, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Share upon request

REFERENCES:
- [Result] Tan SJ, Zhou F, Yui WK, Chen QY, Lin ZL, Hu RY, Gao T, Li N. Fast track programmes vs. traditional care in laparoscopic colorectal surgery: a meta-analysis of randomized controlled trials. Hepatogastroenterology. 2014 Jan-Feb;61(129):79-84. PMID 24895798